CLINICAL TRIAL: NCT02785146
Title: Adjuvant Chemotherapy Combined With Huaier Granule for Treating High-risk Stage II, Stage III Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Qidong Gaitianli Medicines Co., Ltd (Industry)
Responsible Party: Principal Investigator, Xiaojian Wu, Prof., Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: zsly Huaier-1
Record Dates: First submitted 2016-05-19; First posted 2016-05-27 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
Keywords: Huaier Granule; After radical surgery; Prevention of recurrence and metastasis; Efficacy and safety
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — huaier; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mFOLFOX6 + Huaier Granule (Experimental): Twelve cycles of mFOLFOX6 (oxaliplatin, 85 mg/m²; calcium folinate, 400 mg/m²; 5-fluorouracil, 2800 mg/m²). Patients will be treated with chemotherapy every 2 weeks (+/- 2 days ). Huaier Granule will be administrated from the first cycle of chemotherapy until 48 weeks after surgery or until study termination. Huaier Granule is continuously taken three times per day, 20g per time.
  Interventions: Drug: Huaier Granule; Drug: Oxaliplatin; Drug: Calcium folinate; Drug: 5-fluorouracil
- mFOLFOX6 (Active Comparator): Twelve cycles of mFOLFOX6 (oxaliplatin, 85 mg/m²; calcium folinate, 400 mg/m²; 5-fluorouracil, 2800 mg/m²). Patients will be treated with chemotherapy every 2 weeks (+/- 2 days ).
  Interventions: Drug: Oxaliplatin; Drug: Calcium folinate; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: Huaier Granule — Huaier Granule is continuously taken three times per day, 20g per time.
  Other Names: Huaier
  Arms: mFOLFOX6 + Huaier Granule
Drug: Oxaliplatin — 85 mg/m², ivdrip, D1
Drug: Calcium folinate — Calcium folinate 400 mg/m², ivdrip, D1; or calcium levofolinate, 200 mg/m², ivdrip, D1
  Other Names: Calcium levofolinate
Drug: 5-fluorouracil — 400 mg/m², iv, D1; and 2400mg/m², civ, 48h

SUMMARY:
A randomized, paralleled control clinical study investigating Huaier Granule for prevention of recurrence and metastasis of colorectal cancer after radical surgery, to evaluate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* The subjects volunteer to sign the informed consent
* Aged: 18 to 75 years old
* Colorectal cancer (AJCC-TNM, high-risk Stage II and Stage III)
* The diagnosis and colorectal cancer has been confirmed by pathological examination after radical surgery
* The liver and kidney function satisfies the following conditions within 15 days after surgery (excluding day 15): aspartate aminotransferase (AST), glutamic-oxalacetic transaminase (ALT), alkaline phosphatase (ALP)< 2 upper limit of normal (ULN), total bilirubin ≤ 1.5 ULN, serum creatinine < 1.5 ULN; normal coagulation function
* Other laboratory tests meet the following requirements within 15 days after surgery (excluding day 15): white blood cells count ≥ 3.0×109/L, absolute neutrophil count ≥ 1.5×109/L, platelet count ≥ 100×109/L
* ECOG：0-2 points
* No other previous history of malignancy.

Exclusion Criteria:

* Multiple primary cancer
* Not recover from the colorectal surgery
* Presence of organ, bone, or skin metastases
* Pregnant or lactating women
* Those with active bleeding due to various reasons
* Those with HIV infection or AIDS-associated diseases
* Those with severe acute and chronic diseases
* Those with severe diabetes
* Those with serious infectious diseases
* Those who can not take drugs by oral route
* Drug abusers or those with psychological or mental diseases that may interfere with study compliance
* Conditions that are considered not suitable for this study investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 1 year
  DFS was defined as the date of definitive surgery until the date of recurrence, metastasis, appearance of a second primary tumor, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  OS was defined as the date of definitive surgery until the date of death or the last follow-up.
Relapse-free survival (RFS) | 5 years
  RFS was defined as the date of definitive surgery until the date of recurrence or death from any cause.
Metastasis-free survival (MFS) | 5 years
  MFS was defined as the date of definitive surgery until the date of metastasis or death from any cause.

OTHER OUTCOMES:
The effects of Huaier Granule on adverse events of adjuvant chemotherapy. | 6 months
  The adverse events were evaluated every 2 weeks; Eastern Cooperative Oncology Group(ECOG) scores, imaging assessment and related biochemical indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojian Wu, Ph.D., Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The investigators would like to share the data to the Participating units.

REFERENCES:
- [Result] Zhang N, Kong X, Yan S, Yuan C, Yang Q. Huaier aqueous extract inhibits proliferation of breast cancer cells by inducing apoptosis. Cancer Sci. 2010 Nov;101(11):2375-83. doi: 10.1111/j.1349-7006.2010.01680.x. PMID 20718753
- [Result] Wang X, Zhang N, Huo Q, Yang Q. Anti-angiogenic and antitumor activities of Huaier aqueous extract. Oncol Rep. 2012 Oct;28(4):1167-75. doi: 10.3892/or.2012.1961. Epub 2012 Aug 8. PMID 22895629
- [Result] Zhang T, Wang K, Zhang J, Wang X, Chen Z, Ni C, Qiu F, Huang J. Huaier aqueous extract inhibits colorectal cancer stem cell growth partially via downregulation of the Wnt/beta-catenin pathway. Oncol Lett. 2013 Apr;5(4):1171-1176. doi: 10.3892/ol.2013.1145. Epub 2013 Jan 21. PMID 23599758
- [Result] Wang X, Zhang N, Huo Q, Sun M, Dong L, Zhang Y, Xu G, Yang Q. Huaier aqueous extract inhibits stem-like characteristics of MCF7 breast cancer cells via inactivation of hedgehog pathway. Tumour Biol. 2014 Nov;35(11):10805-13. doi: 10.1007/s13277-014-2390-2. Epub 2014 Jul 31. PMID 25077927